CLINICAL TRIAL: NCT05870631
Title: Immunogenicity and Safety of Adsorbed Diphtheria, Tetanus, Acellular Pertussis Combined Vaccine or Adsorbed Diphtheria Tetanus Combined Vaccine in 6 Years Old Children#a Randomized, Controlled Clinical Study
Brief Title: Immunogenicity and Safety of DTaP or DT Vaccine in 6 Year Old Children ( DTaP/DT )
Acronym: DTaP/DT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Provincial Center for Disease Control and Prevention (Other Government)
Collaborators: China National Biotec Group Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DTaP/DT-2023-02
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Vaccine Reaction
Keywords: immunogenicity，safety，DTap，DT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group with DTap vaccination produced by Chendu Institute of Biological Products Co., Ltd
  Interventions: Biological: vaccinate with DTaP
- Group B (Experimental): Group with DT vaccination
  Interventions: Biological: vaccinate with DT

INTERVENTIONS:
Biological: vaccinate with DTaP — vaccinate with DTaP
  Arms: Group A
Biological: vaccinate with DT — vaccinate with DT
  Arms: Group B

SUMMARY:
This study is to evaluate the immunogenicity and safety of DTaP or DT given in children aged 6 years.

DETAILED DESCRIPTION:
A phase 4 trial was conducted in Zhejiang Province aimed to evaluate the immunogenicity and safety of DTaP or DT in children aged 6 years. DTaP and DT are produced by Chengdu Institute of Biological Products Co., Ltd. Participants will be recruited and randomly divided into two groups to receive DTaP or DT in 1:1 ratio. Two blood samples were taken on Day 0 (pre-vaccination) and Day 28~42 (after-vaccination) for test antibody against pertussis, diphtheria and tetanus. Adverse events and serious adverse events were actively collected by staff within 28 days of vaccination.

ELIGIBILITY:
Inclusion Criteria:

* 1. Participants aged ≥ 6 on the day of enrollment; 2. Informed consent should be signed and dated by the participants; 3. The participant's legal guardian is able to attend all planned follow-up visits and comply with all study procedures; 4. The participants have received 4 doses of acellular TDap vaccine and have not received any immunization agents related to diphtheria, tetanus, and pertussis in the past 3 years; 5. The participant has no diease history of pertussis, diphtheria or tetanus; 6. ≥ 14 days interval between the last vaccination; 7. Body temperature was ≤37.3℃.

Exclusion Criteria:

* 1、Being allergic to any component of vaccines ； 2、A history of severe allergic reactions to any vaccine (for example acute allergic reaction, angioneurotic edema, dyspnea, etc）； 3、Having a history or family history of convulsions, encephalopathy, psychosis, uncontrolled epilepsy and other progressive neurological diseases; 4、Participants are suffering from immunodeficiency, receiving immunosuppressant therapy (oral steroid hormones) during treatment for malignancy, or having low immunity due to HIV, or having congenital immune disorders in close family members; 5、Injection of non-specific immunoglobulin within 1 month before enrollment; 6、Participants are suffering from acute febrile diseases and infectious diseases; 7、A history of clearly diagnosed thrombocytopenia or other clotting disorders that may contraindicate subcutaneous injection; 8、Participants with severe chronic diseases or acute episodes of chronic diseases; 9、Participants with infectious, suppurative and allergic skin diseases; 10、Other Participants whose physical conditions, as determined by the investigator, are not suitable for inclusion in clinical studies.

Ages: 72 Months to 84 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rates of the vaccination | 28-42 days after the dose of DTaP or DT
  Defined as any positive antibody response against pertussis，diphtheria，tetanus in children who were seronegative prior to the vaccination, or at least a fourfold increase in antibody levels against pertussis for children who had pre-existing positive antibodies
Seropositive rates after the vaccination | 28-42 days after the dose of DTaP or DT
  The percentage of participants with positive antibody against pertussis，diphtheria and tetanus.

SECONDARY OUTCOMES:
Safety of the DTaP or DT vaccine immunization | 28 days after the vaccination
  The occurrence of adverse events for vaccination administered at age 6 using DTaP or DT
Geometric mean antibody concentrations before the vaccination | before the dose of DTaP or DT
  The GMC against pertussis，diphtheria and tetanus
Geometric mean antibody concentrations after the vaccination | 28-42 days after the dose of DTaP or DT
  The GMC against pertussis，diphtheria and tetanus

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fuyang Center for Disease Control and Prevention, Hangzhou, Zhejiang
  - Tongxiang Center for Disease Control and Prevention, Jiaxing, Zhejiang

IPD SHARING:
Plan to Share IPD: No